CLINICAL TRIAL: NCT05559853
Title: Development of a Clinical CEST MR Fingerprinting Method for Treatment Response Assessment in Brain Metastases
Brief Title: Developing a New MRI Technique to Understand Changes in Brain Tumors After Treatment
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 22-191
Record Dates: First submitted 2022-09-22; First posted 2022-09-29 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Brain Metastases; Brain Metastases, Adult; Metastatic Brain Tumor; Metastatic Brain Cancer
Keywords: Brain Metastases; Healthy Volunteers; metastatic brain tumor; metastatic brain cancer; Brain Metastases, Adult; MRI; untreated brain metastasis; CEST-MRF; chemical exchange saturation transfer magnetic resonance fingerprinting; 22-191; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Participants with Brain Metastases: Participants will have at least one untreated brain metastasis > 1cm
  Interventions: Diagnostic Test: CEST-MRF
- Healthy participants: Participants will have no known cancer diagnosis. Volunteers enrolled on this protocol may undergo multiple MRI examinations periodically for studies of reproducibility.
  Interventions: Diagnostic Test: CEST-MRF

INTERVENTIONS:
Diagnostic Test: CEST-MRF — CEST-MRF enables accurate quantification of both proton exchange rates and volume fractions in a fraction of the time required by conventional pulse sequences will be developed and optimized.
  Other Names: chemical exchange saturation transfer magnetic resonance fingerprinting method

SUMMARY:
The purpose of this study is to develop and test a new magnetic resonance imaging (MRI) technique to see if it can be used to tell the difference between tumor growth from worsening of cancer and growth from the effects of treatment in participants who have brain tumors treated with radiation therapy called stereotactic radiosurgery (SRS).

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers [for Study Aim 1 (SA1) and Study Aim 2 (SA2)] will be entered into the study if they meet the following criteria:

* Age ≥ 18 years
* Able to understand and give informed consent
* No known cancer diagnosis

Patients [for Study Aim 1 (SA1)] will be entered into the study if they meet the following criteria:

* Age ≥ 18 years
* Able to understand and give informed consent
* At least one untreated brain metastasis > 1cm (e.g., an enhancing lesion in the brain of a patient with known systemic cancer determined likely to represent metastasis by neuroradiologist)

Patients [for Study Aim 3 (SA3)] will be entered into the study if they meet the following criteria:

* Age ≥ 18 years
* Able to understand and give informed consent
* At least one untreated brain metastasis > 1cm (e.g., an enhancing lesion in the brain of a patient with known systemic cancer determined likely to represent metastasis by neuroradiologist)
* Planned SRS treatment

Exclusion Criteria:

Healthy volunteers (SA1 & SA2) and patients (SA1 & SA3) exclusion criteria:

* Pregnant or breastfeeding women
* Pre-existing medical conditions, including the likelihood of developing seizures or claustrophobic reactions, and any greater than normal potential for cardiac arrest
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study investigators will discuss participant potentially eligible for research participation within their interdisciplinary brain metastasis disease management team. These potential participants will then be contacted by their treating physician or investigator team. Study investigators will prioritize consenting participants who are planned to undergo SRS and, when possible, will attempt to coordinate the research scan with their clinically necessary MRI scans to minimize time and disruption for the participant.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2027-09-22 (Estimated); Study Completion 2027-09-22 (Estimated)

PRIMARY OUTCOMES:
Change of Rapid chemical exchange saturation transfer (CEST) imaging with magnetic resonance fingerprinting (MRF)/CEST-MRF parameters with and without motion | Up to 3 years
  Develop a rapid and robust 3D CEST-MRF pulse sequence for clinical scanners using our preclinical CEST-MRF pulse sequence as a basis by evaluating the changes of the 6 CEST-MRF parameters with and without motion. These parameters include the water T1 and T2 relaxation (T1w,T2w), amide exchange rate (ksw) and volume fraction (fs) and the semi-solid exchange rate (kssw) and volume fraction (fss).

SECONDARY OUTCOMES:
Create CEST-MRF parameter maps | Up to 3 years
  Develop an MRI physics-guided artificial intelligence approach to improve acquisition and reconstruction of multiparametric data
Measure longitudinal changes in CEST-MRF after SRS | Up to 3 years
  Evaluate CEST-MRF changes before and after radiation therapy to assess potential role as predictive imaging biomarker for brain metastases

CONTACTS AND LOCATIONS:
Overall Officials: Ouri Cohen, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org